CLINICAL TRIAL: NCT02732769
Title: Clinical Evaluation of the Treatment of Intellectual Metastases by Radiosurgery Gamma Knife by Means of a Support System by Mask.
Acronym: Mask
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2015-40; 2015-A01673-46 (Registry Identifier: Ansm)
Record Dates: First submitted 2016-03-30; First posted 2016-04-11 (Estimated); Last update posted 2018-10-03 (Actual); Status verified 2016-04

CONDITIONS: Lung Cancer; Brain Metastases
MeSH Terms: conditions — Lung Neoplasms; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group treated by radiosurgery with stereotaxic frame (Active Comparator): Subjects will receive a radiosurgery during a brief hospitalization by LeksellGammaKnifePerfexion® (LGKP)
  Interventions: Device: GammaKnifePerfexion®; Device: MRI
- Group treated by radiosurgery with the thermoformed mask (Experimental): Subjects will receive a radiosurgery with thermoformed mask during a brief hospitalization by GammaKnifeICON® (GKI) with Efficast®
  Interventions: Device: GammaKnifeIcon®; Device: Efficast®; Device: MRI

INTERVENTIONS:
Device: GammaKnifePerfexion® — neurosurgery
  Arms: Group treated by radiosurgery with stereotaxic frame
Device: GammaKnifeIcon® — neurosurgery
  Arms: Group treated by radiosurgery with the thermoformed mask
Device: Efficast® — Thermoformed mask
  Arms: Group treated by radiosurgery with the thermoformed mask
Device: MRI

SUMMARY:
the Mask fixation isn't a new solution for the immobilization of the patient's head and has been used in current practice for long years.

This trial is attempting to compare these two technical possibilities of head fixation by mask or by stereotaxic frame. The primary goal is to evaluate the comfort for the patient and specifically for each step of the procedure. It will also evaluate other parameters such as the effectiveness of these two strategies and tolerance.The expected benefit is an improvement of the comfort for the patients.

ELIGIBILITY:
Inclusion Criteria:

* Subject bearing of one to five intellectual metastases of lung origin at the time of the indication of the radiosurgery
* Subject requiring a radiosurgical treatment with LGK

Exclusion Criteria:

* Subject having hurts of the brainstem or para-optics
* Pregnant women or in feeding period
* Subject having received previously a whole brain radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-07-27 (Actual); Study Completion 2018-03-21 (Actual)

PRIMARY OUTCOMES:
Evaluation of pain during the hospitalization (3 days) | 12 months
  Questionary (numeric pain intensity scale)

SECONDARY OUTCOMES:
Evaluation of tumor control at 3 months | 12 months
  No increase of volume greater than 50% on the MRI
Evaluation of tumor control at 6 months | 12 months
  No increase of volume greater than 50% on the MRI
Occurrence of clinical side effects | 12 months
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: DESALBRES, Study Director — ASSISTANCE PUBLIQUE HÔPITAUX DE MARSEILLE
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No